CLINICAL TRIAL: NCT04186832
Title: Feasibility of Monitoring Step Count as a Measure of Physical Activity in Patients With Newly Diagnosed Glioma Patients Undergoing Radiation Therapy
Brief Title: Step Count Monitoring as a Measure of Physical Activity in Patients With Newly Diagnosed Glioma Undergoing Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0564; NCI-2019-06739 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0564 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-20; First posted 2019-12-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Radiation Therapy Patient
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (pedometer) (Active Comparator): Patients wear a pedometer for step count monitoring over 6 weeks.
  Interventions: Device: Pedometer; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (FitBit) (Experimental): Patients wear a FitBit for step count monitoring over 6 weeks.
  Interventions: Device: FitBit; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Device: FitBit — Wear FitBit
  Arms: Group II (FitBit)
Device: Pedometer — Wear pedometer
  Arms: Group I (pedometer)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the feasibility of monitoring step count as a measure of physical activity in patients with newly diagnosed glioma undergoing radiation therapy. Physical activity measured by step count may help to improve the quality of life and symptoms for patients with newly diagnosed glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of monitoring step count as a measure of physical activity in patients with newly diagnosed glioma undergoing radiation therapy (RT) at MD Anderson Cancer Center (MDACC).

SECONDARY OBJECTIVE:

I. Estimate the effects of physical activity as measured by step count on cognition, fatigue, anxiety and depression scores and assess differences between groups.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients wear a pedometer for step count monitoring over 6 weeks.

GROUP II: Patients wear a FitBit for step count monitoring over 6 weeks.

After completion of study, patients are followed up at 3 and 6 months after completing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a glioma and going to receive at least 4 weeks of RT at MDACC at the Texas Medical Center campus with at least 20 fractions
* Karnofsky performance status (KPS) of 70 or above
* Wearable activity tracker (WAT) - naive
* Able to read and speak English
* Able to provide informed consent
* Access to a smartphone
* Access to Wi-Fi

Exclusion Criteria:

* Cognitive and/or major sensory deficits that would impede the completion of assessment instruments as deemed by the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Consent rate | Up to 6 months after completing radiation therapy
  Feasibility will be assessed by the consent rate. Will calculate the rates, frequencies, and 90% confidence intervals (CIs) of the proportions by group and in total, as well as for the differences between intervention groups, as applicable.
Fitbit adherence rate | Up to 6 weeks
  Feasibility will be assessed by treatment group (Fitbit) adherence rate. Intervention adherence is defined as wearing the Fitbit for a total of at least 340 hours across the 6-week intervention period. Will calculate the rates, frequencies, and 90% CIs of the proportions by group and in total, as well as for the differences between intervention groups, as applicable.
Retention rate | Up to 6 months
  Feasibility will be assessed by the retention rate. Retention will be defined by the completion of assessments, by the end of the intervention (6 weeks from baseline) in each group. Will calculate the rates, frequencies, and 90% CIs of the proportions by group and in total, as well as for the differences between intervention groups, as applicable.
Satisfaction/acceptability rate questionnaire | Up to 6 months
  Will evaluate the satisfaction/acceptability rate in both FitBit and pedometer groups. Will calculate the rates, frequencies, and 90% CIs of the proportions by group and in total, as well as for the differences between intervention groups, as applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei S Weathers, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org